CLINICAL TRIAL: NCT02778204
Title: Phase I Safety and Pharmacokinetic Study of Maraviroc in HIV-1-Exposed Infants at Risk of Acquiring HIV-1 Infection
Brief Title: Evaluating the Safety and Pharmacokinetics of Maraviroc in HIV-1-Exposed Infants at Risk of Acquiring HIV-1 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); ViiV Healthcare (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT 2007; 20734 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections
Keywords: Vertical HIV exposure; Neonates; Maraviroc
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Stratum 1A (Experimental): Infants in this cohort received a single dose of 8 mg/kg maraviroc solution within 3 days of birth and at Week 1 (7-14 days) of life; without in utero exposure to maternal efavirenz.
  Interventions: Drug: Maraviroc
- Cohort 1 Stratum 1B (Experimental): Infants in this cohort received a single dose of 8 mg/kg maraviroc solution within 3 days of birth and at Week 1 (7-14 days) of life; with in utero exposure to maternal efavirenz.
  Interventions: Drug: Maraviroc
- Cohort 2 Stratum 2A (Experimental): Infants in this cohort received 8 mg/kg maraviroc solution twice daily starting within 3 days of birth and continuing up to Week 6 (35-42) days of life; without in utero or breast milk exposure to maternal efavirenz.
  Interventions: Drug: Maraviroc
- Cohort 2 Stratum 2B (Experimental): Infants in this cohort received 8 mg/kg maraviroc solution twice daily starting within 3 days of birth and continuing up to Week 6 (35-42) days of life; with in utero and breast milk exposure to maternal efavirenz
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — 8 mg/kg oral solution as a single dose.
  Arms: Cohort 1 Stratum 1A; Cohort 1 Stratum 1B
Drug: Maraviroc — 8 mg/kg oral solution given twice daily.
  Arms: Cohort 2 Stratum 2A; Cohort 2 Stratum 2B

SUMMARY:
This study aimed to evaluate the safety, tolerability, and pharmacokinetics of maraviroc in infants at risk for mother-to-child HIV transmission, and to determine an appropriate dose of maraviroc during the first six weeks of life.

DETAILED DESCRIPTION:
Maraviroc is a C-C Chemokine Receptor 5 (CCR5) receptor antagonist used to treat HIV infection in adults. Adding maraviroc to a standard of care prophylaxis regimen may also reduce the risk of perinatal transmission of HIV. The purpose of this study was to evaluate the safety, tolerability, and pharmacokinetics of maraviroc in HIV-1-exposed infants at risk for mother-to-child HIV transmission. This study also aimed to determine an appropriate dose of maraviroc during the first six weeks of life.

The study allowed up to 72 mother-infant pairs in two cohorts to achieve a target of 36 evaluable infants receiving the final recommended dose of maraviroc. Because maraviroc interacts with the antiretroviral drug efavirenz (EFV) in adults, infants in this study were stratified within the cohorts based on their exposure to maternal EFV. Cohort 1 was stratified by in utero exposure to maternal EFV, with infants in both strata receiving a single dose of maraviroc solution within three days of birth and another single dose at Week 1 of life. Stratum 1A included infants without in utero exposure to maternal EFV during the eight weeks immediately before delivery. Stratum 1B included infants with in utero exposure to maternal EFV for a minimum of two weeks immediately before delivery.

Cohort 2 was stratified by exposure to maternal EFV after birth, with infants in both strata receiving maraviroc oral solution twice daily starting within three days of birth and continuing for up to 42 days. Based on evaluation of the Cohort 1 data, the initial daily dose of maraviroc oral solution to be administered in Cohort 2 was 8 mg/kg dose given twice daily. Stratum 2A included infants without any exposure to maternal EFV either in utero during the eight weeks immediately before delivery or while breastfeeding. Stratum 2B included breastfeeding infants with exposure to maternal EFV both in utero and after birth while breastfeeding, for a minimum of 2 weeks immediately before delivery and while breastfeeding.

Participants attended an entry visit within three days after the infant's birth. Participants attended five to six study visits through Week 16. Visits included medical history reviews, physical examinations, blood collection from the mother and/or infant, HIV testing, and adherence counseling.

ELIGIBILITY:
Inclusion Criteria:

* Mother was of legal age to provide independent informed consent for research participation and was willing and able to provide written informed consent for her and her infant's participation in this study.
* Mother had confirmed HIV-1 infection based on testing of two samples collected at different time points. More information on this criterion can be found in the protocol.
* At entry, infant met EFV exposure requirements, based on mother's report and confirmed by medical records if available, as follows:

  * For Cohort 1, Stratum 1A: Infant born to a mother who did not receive EFV during the eight weeks immediately prior to delivery. Note: Breastfeeding and formula feeding infants were eligible for this stratum.
  * For Cohort 1, Stratum 1B: Infant born to a mother who received EFV for a minimum of two weeks immediately prior to delivery. Note: Breastfeeding and formula feeding infants were eligible for this stratum.
  * For Cohort 2, Stratum 2A: Infants born to a mother who did not receive EFV during the eight weeks immediately prior to delivery and if breastfeeding, mother was not receiving maternal EFV. Note: Breastfeeding and formula feeding infants were eligible for this stratum.
  * For Cohort 2, Stratum 2B: Breastfeeding infants born to a mother who received EFV for a minimum of two weeks immediately prior to delivery, intended to breastfeed for a minimum of six weeks and continued to receive maternal EFV while breastfeeding. Note: Only breastfeeding infants were eligible for this stratum.
* At birth, infant's estimated gestational age was at least 37 weeks. Note: If gestational age at birth is not documented in the infant's available birth records, study staff may assess gestational age at the earliest possible opportunity during the screening period and use this assessment for purposes of eligibility determination.
* At birth, infant's weight was at least 2 kg. Note: If weight at birth is not documented in the infant's available birth records, study staff may assess infant weight at the earliest possible opportunity during the screening period and use this assessment for purposes of eligibility determination.
* At entry, infant was less than or equal to 3 days old.
* At entry, infant had the following lab values:

  * Grade 0 alanine transaminase (ALT) (normal)
  * Less than or equal to Grade 1 aspartate aminotransferase (AST) and total bilirubin
  * Less than or equal to Grade 2 hemoglobin, white blood cell counts, platelet counts
* At entry, infant had initiated antiretroviral prophylaxis that did not include a potent CYP3A4 inhibitor or inducer. See the protocol for more information.
* At entry, infant was assessed by the site investigator or designee as generally healthy based on review of available medical records, other available medical history information, and physical examination findings.
* Born after singleton delivery (not after multiple birth).

Exclusion Criteria:

* Infant had any other condition that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives; for example, severe congenital malformation, other medical condition, or clinically significant finding from physical examination.
* At entry, any positive infant HIV nucleic acid test result (results are not required to be available prior to entry but any positive results obtained prior to entry are exclusionary).
* At entry, infant or breastfeeding mother was receiving any disallowed medication listed in the protocol.
* Mother received maraviroc during pregnancy.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, MD, Study Chair — Boston University School of Medicine/Boston Medical Center
Locations (9):
- United States (5):
  - Usc La Nichd Crs, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
- Kenya Medical Research Institute / Walter Reed Project Clinical Research Center, Kericho CRS, Kericho, Kenya
- South Africa (2):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Umlazi CRS, Durban, KwaZulu-Natal
- Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi, Thailand

REFERENCES:
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, dated July 2017 — https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual occurred between June 2017 and July 2019 in Kenya, Thailand, South Africa, and the United States at 9 different medical clinic sites. Pregnant mothers were screened and subsequently enrolled for 1 day at the same day their newborn infants were enrolled (within 3 days of life).
Pre-assignment Details: The sample size of the study (47) represents the infants enrolled. As multiple births are disallowed in the study, this also represents the total mother-infant pairs.
Period: Overall Study
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Started | 8 | 7 | 16 | 16
Completed | 6 | 7 | 12 | 12
Not Completed | 2 | 0 | 4 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Eligibility Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all infants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B | Total
Number analyzed (Participants) | 8 | 7 | 16 | 16 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: days] — This is the Infant age at baseline.
  days
    Mean (Standard Deviation) | 1.5 [1 to 2] | 0 [0 to 1] | 1 [0 to 2] | 2 [2 to 3] | 2 [1 to 2]
Age, Continuous [Median (Inter-Quartile Range); unit: years] — This is the Maternal Age at baseline.
  years | 29.5 [29 to 37] | 26 [24 to 39] | 32 [26.5 to 36] | 32 [27.5 to 37.5] | 31 [26 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 7 | 7 | 23
  Male | 3 | 3 | 9 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 0 | 5
  Not Hispanic or Latino | 5 | 7 | 14 | 16 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 10 | 16 | 38
  White | 3 | 0 | 3 | 0 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 0 | 13 | 0 | 20
  South Africa | 1 | 7 | 0 | 14 | 22
  Thailand | 0 | 0 | 3 | 0 | 3
  Kenya | 0 | 0 | 0 | 2 | 2
Birth Weight [Median (Inter-Quartile Range); unit: kilograms] | 3.2 [2.8 to 3.5] | 3.4 [2.9 to 3.64] | 3.0 [2.9 to 3.19] | 3.0 [2.8 to 3.16] | 3.05 [2.9 to 3.4]
Birth Length [Median (Inter-Quartile Range); unit: centimeters] | 50.0 [49.0 to 51.25] | 50.0 [48.5 to 51.0] | 49.0 [49.0 to 50.5] | 48.5 [47.5 to 50.45] | 49.0 [48.0 to 51.0]
Gestational Age [Median (Inter-Quartile Range); unit: weeks] | 38.5 [38.0 to 39.5] | 39.0 [38.0 to 39.0] | 39.0 [38.0 to 39.5] | 40.0 [39.0 to 40.5] | 39.0 [38.0 to 40.0]
APGAR at 1 minute [Median (Inter-Quartile Range); unit: units on a scale] — APGAR Score ranges from 1-10, with 1 being the worst and 10 being the best.
  units on a scale | 9.0 [9.0 to 9.0] | 8.0 [8.0 to 8.0] | 8.5 [8.0 to 9.0] | 9.0 [8.0 to 9.0] | 9.0 [8.0 to 9.0]
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: ukat/L] | 0.2 [0.1 to 0.23] | 0.2 [0.2 to 0.28] | 0.2 [0.1 to 0.25] | 0.2 [0.1 to 0.24] | 0.2 [0.1 to 0.25]
Aspartate Aminotransferase (AST) [Median (Inter-Quartile Range); unit: ukat/L] | 0.7 [0.5 to 0.91] | 1.1 [0.9 to 3.46] | 0.9 [0.6 to 1.08] | 1.0 [0.7 to 1.27] | 0.9 [0.7 to 1.15]
Total Bilirubin [Median (Inter-Quartile Range); unit: umol/L] | 39.3 [30.8 to 74.8] | 44.0 [25.0 to 49.0] | 76.1 [41.0 to 129.1] | 75.3 [41.6 to 105.3] | 50.7 [35.9 to 99.2]
Creatinine [Median (Inter-Quartile Range); unit: umol/L] | 70.7 [54.4 to 78.7] | 62.0 [54.0 to 63.0] | 61.9 [49.5 to 70.7] | 69.0 [44.0 to 73.0] | 66 [49.5 to 72.0]
Platelets [Median (Inter-Quartile Range); unit: 10^9 platelets/L] | 274.0 [247.0 to 335.5] | 297.0 [272.0 to 380.0] | 252.5 [161.5 to 307.5] | 311.0 [261.0 to 383.5] | 289.0 [241.0 to 360.0]
Hemoglobin [Median (Inter-Quartile Range); unit: g/L] | 163.0 [158.5 to 166.5] | 178.0 [171.0 to 216.0] | 166.5 [152.5 to 174.0] | 179.0 [165.5 to 205.5] | 170.0 [161.0 to 194.0]
White Blood Cell Count (WBC) [Median (Inter-Quartile Range); unit: 10^9 cells/L] | 14.6 [12.0 to 19.65] | 17.3 [12.9 to 19.3] | 15.5 [12.2 to 20.0] | 12.6 [10.6 to 15.7] | 14.6 [11.3 to 17.4]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Failing to Meet Safety Endpoint Related to Maraviroc for Dose-Finding
Description: Percentage (%) of failure and Clopper-Pearson 95% Confidence Interval (CI). Failure is defined as having: Any life threatening adverse event (AE), including death, assessed as at least possibly related to the study drug, AEs of Grade 3 or higher judged by the Core Protocol Team to be probably or definitely related to the study drug, or that result in permanent discontinuation of study drug due to an AE, judged by Core Protocol Team to be at least possibly related to study drug
Time Frame: Cohort 1: Measured from first dose of maraviroc to 7 Day Post Dose Visit (up to 25 days). Cohort 2: Measured from first dose of maraviroc to Week 6 Visit (up to 42 days).
Population: Safety-evaluable population are those who were taking maraviroc for the expected time-frame (Cohort 1: through 7 day post-dose visit, Cohort 2: Through week 6)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 12 | 12
percentage of participants | 0 [0 to 45.9] | 0 [0 to 41.0] | 0 [0 to 26.5] | 0 [0 to 26.5]

2. Primary Outcome: Percentage of Participants Failing to Meet Safety Endpoint Related to Maraviroc for Analysis
Description: Percentage (%) of failure and Clopper-Pearson 95% CI. Failure is defined as: Any life threatening AE, including death, assessed as at least possibly related to the study drug, AEs of Grade 3 or higher judged by the Core Protocol Team to be probably or definitely related to the study drug, or that result in permanent discontinuation of study drug due to an AE, judged by Core Protocol Team to be at least possibly related to study drug
Time Frame: Measured from first dose of maraviroc to Week 6 Visit (up to 42 days)
Population: Analysis Endpoint includes all treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 8 | 7 | 16 | 16
percentage of participants | 0 [0 to 36.9] | 0 [0 to 41.0] | 0 [0 to 20.6] | 0 [0 to 20.6]

3. Primary Outcome: Number of Participants Failing to Meet PK Target
Description: Number of failures. The pharmacokinetic (PK) target is Average Concentration (Cavg) greater than or equal to 75 ng/mL (based on a dose interval of every 12 hours). Failure is defined as Cavg <75 ng/mL at each intensive PK visit.
  For Cohort 1:
  For the Entry Visit, PK samples were drawn at: pre-dose and at 1-2, 4-8, 11-13, 20-24, and 48-72 hours post-dose. For the Week 1 Visit, PK samples were drawn at: pre-dose and 1-2 and 22-26 hours post-dose.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: Cohort 1: Measured at Entry (First visit) and Week 1 Visit (Second visit). Cohort 2: Measured at Week 1 (First visit) and Week 4 Visit (Second visit).
Population: Analysis population included dose-finding evaluable participants with intensive pharmacokinetic (PK) results.
  In Cohort 1 Stratum 1A and 1B at the week 1 visit (Second Visit), only 3 PK sample were drawn (pre-dose, 1-2 hours post-dose, and 22-26 hours post-dose). Maraviroc was only measurable (above assay limit) at 1 time point (1-2 hours post-dose). Therefore, AUC (hence Cavg) could not be estimated with non-compartmental methods from only 1 concentration and thus the number analyzed was 0.
Measure: Number; unit: participants
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 13 | 12
participants
  First Visit | 0 | 0 | 3 | 4
  Second Visit: number analyzed (Participants) | 0 | 0 | 13 | 12
  Second Visit |  |  | 4 | 5

4. Primary Outcome: Pharmacokinetic (PK) Parameter: Average Concentration (Cavg)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (Phoenix 64, WinNonlin, Pharsight Corp., Mountain View, CA). Cavg was determined as the area-under-the-curve (AUC) divided by the dose interval, tau (τ) of every 12 hours.
  For Cohort 1:
  For the Entry Visit, PK samples were drawn at: pre-dose and at 1-2, 4-8, 11-13, 20-24, and 48-72 hours post-dose. For the Week 1 Visit, PK samples were drawn at: pre-dose and 1-2 and 22-26 hours post-dose.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: Cohort 1: Measured at Entry and Week 1 Visit. Cohort 2: Measured at Week 1 and Week 4 Visit
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 13 | 12
ng/mL
  First Visit | 190.47 [93.54 to 1278.62] | 375.47 [110.40 to 684.84] | 152.24 [19.75 to 565.68] | 124.67 [17.07 to 550.86]
  Second Visit: number analyzed (Participants) | 0 | 0 | 13 | 12
  Second Visit |  |  | 93.58 [32.92 to 488.21] | 101.39 [42.65 to 351.19]

5. Primary Outcome: Pharmacokinetic (PK) Parameter: Area-under-the-curve (AUC)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (Phoenix 64, WinNonlin, Pharsight Corp., Mountain View, CA). For Cohort 1 (single doses), area-under-the-curve (AUC) was determined from time zero to infinity. For Cohort 2 (at steady-state), area-under-the-curve (AUC) was determined from time pre-dose to tau (12 hours).
  For Cohort 1:
  For the Entry Visit, PK samples were drawn at: pre-dose and at 1-2, 4-8, 11-13, 20-24, and 48-72 hours post-dose. For the Week 1 Visit, PK samples were drawn at: pre-dose and 1-2 and 22-26 hours post-dose.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 13 | 12
ng*hr/mL
  First Visit | 2285.68 [1122.53 to 15343.42] | 4506.17 [1325.02 to 8218.03] | 1826.87 [236.96 to 6788.18] | 1496.05 [204.89 to 6610.35]
  Second Visit: number analyzed (Participants) | 0 | 0 | 13 | 12
  Second Visit |  |  | 1122.99 [395.01 to 5858.51] | 1216.62 [511.85 to 4214.34]

6. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Concentration (Cmax)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles. Cmax was the observed highest concentration.
  For Cohort 1:
  For the Entry Visit, PK samples were drawn at: pre-dose and at 1-2, 4-8, 11-13, 20-24, and 48-72 hours post-dose. For the Week 1 Visit, PK samples were drawn at: pre-dose and 1-2 and 22-26 hours post-dose.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: as for outcome 3
Population: Analysis population included dose-finding evaluable participants with intensive pharmacokinetic (PK) results.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 13 | 12
ng/mL
  First Visit | 227.3 [29.9 to 1618.4] | 550.5 [203.8 to 1153] | 256.9 [51.5 to 1468.4] | 308.8 [34.4 to 1273.5]
  Second Visit | 128.9 [22.8 to 296.2] | 163.4 [8.7 to 609.4] | 416.5 [125.1 to 793.4] | 221.8 [76.5 to 738.7]

7. Primary Outcome: Pharmacokinetic (PK) Parameter: Time of Maximum Concentration (Tmax)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles. Tmax was the time at which Cmax, the observed highest concentration, occurred.
  For Cohort 1:
  For the Entry Visit, PK samples were drawn at: pre-dose and at 1-2, 4-8, 11-13, 20-24, and 48-72 hours post-dose. For the Week 1 Visit, PK samples were drawn at: pre-dose and 1-2 and 22-26 hours post-dose.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: as for outcome 3
Population: Analysis population included dose-finding evaluable participants with intensive pharmacokinetic (PK) results.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 13 | 12
hours
  First Visit | 4.68 [1.05 to 12.75] | 1.52 [1.25 to 4.42] | 1.50 [0.83 to 4.00] | 3.00 [1.00 to 6.18]
  Second Visit | 1.18 [1.05 to 1.25] | 1.08 [1.07 to 1.33] | 1.50 [1.00 to 4.00] | 2.19 [0.00 to 11.43]

8. Primary Outcome: Pharmacokinetic (PK) Parameter: Trough Concentration (Ctau)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles. Ctau was the observed concentration at the trough time of 12 hours post-dose with steady-state dosing.
  For Cohort 2:
  For both intensive PK visits, PK samples were drawn at: pre-dose and 1-2, 3-5, 6-8, and 11-13 hours post-dose.
Time Frame: Measured at Week 1 and Week 4 Visit
Population: Analysis population included Cohort 2 dose-finding evaluable participants with intensive pharmacokinetic (PK) results.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 13 | 12
ng/mL
  Week 1 Visit | 27.9 [0 to 138.9] | 23.4 [0 to 824.9]
  Week 4 Visit | 34.4 [0 to 373.1] | 54.9 [8.2 to 233.9]

9. Secondary Outcome: Percentage of Participants Failing to Meet Long-Term Safety Endpoint Related to Maraviroc for Dose-Finding
Description: Percentage (%) of failure and Clopper-Pearson 95% CI. Failure is defined as having: Any life threatening AE, including death, assessed as at least possibly related to the study drug, AEs of Grade 3 or higher judged by the Core Protocol Team to be probably or definitely related to the study drug, or that result in permanent discontinuation of study drug due to an AE, judged by Core Protocol Team to be at least possibly related to study drug
Time Frame: Measured from first dose of maraviroc to Week 16 Visit (up to 140 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 6 | 7 | 12 | 12
percentage of participants | 0 [0 to 45.9] | 0 [0 to 41.0] | 0 [0 to 26.5] | 0 [0 to 26.5]

10. Secondary Outcome: Percentage of Participants Failing to Meet Long-Term Safety Endpoint Related to Maraviroc for Analysis
Description: as for outcome 9
Time Frame: Measured from first dose of maraviroc to Week 16 Visit (up to 140 days)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
Number analyzed (Participants) | 8 | 7 | 16 | 16
percentage of participants | 0 [0 to 36.9] | 0 [0 to 41.0] | 0 [0 to 20.6] | 0 [0 to 20.6]

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Week 16 or premature study discontinuation
Description: All new diagnoses, signs/symptoms and laboratory events of ≥Grade 1 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade, were collected. Adverse events (AE) were graded according to the 246 Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, dated July 2017
Arm/Group | Cohort 1 Stratum 1A | Cohort 1 Stratum 1B | Cohort 2 Stratum 2A | Cohort 2 Stratum 2B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/7 | 4/16 | 2/16
Other Adverse Events (participants affected / at risk) | 7/8 | 7/7 | 15/16 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Stratum 1A (N=8) | Cohort 1 Stratum 1B (N=7) | Cohort 2 Stratum 2A (N=16) | Cohort 2 Stratum 2B (N=16)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Slow response to stimuli (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Stratum 1A (N=8) | Cohort 1 Stratum 1B (N=7) | Cohort 2 Stratum 2A (N=16) | Cohort 2 Stratum 2B (N=16)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Congenital melanocytic naevus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Conjunctival pallor (Eye disorders) | 0 | 1 | 0 | 1
Eye discharge (Eye disorders) | 1 | 1 | 0 | 3
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Orbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Genital candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Ophthalmia neonatorum (Infections and infestations) | 1 | 0 | 1 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 3
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 9 | 4
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 4 | 4 | 11 | 5
Neutrophil count decreased (Investigations) | 0 | 2 | 5 | 7
Weight decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Underweight (Metabolism and nutrition disorders) | 3 | 1 | 4 | 0
Acquired macrocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3 | 2
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 3
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 3
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
As with other Antiretrovirals (ARVs) in young infants, maraviroc PK parameters showed high intra- and inter-participant variability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (4):
  • Study Protocol (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT02778204/Prot_003.pdf
  • Statistical Analysis Plan: Primary Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02778204/SAP_001.pdf
  • Statistical Analysis Plan: PK Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT02778204/SAP_002.pdf
  • Informed Consent Form (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02778204/ICF_000.pdf